CLINICAL TRIAL: NCT06606886
Title: Effects of Hydroxyurea and Metformin in Transfusion Dependent Beta-Thalassemia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUHS-IRB # R-063/24
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Transfusion Dependent Beta-thalassemia
Keywords: Beta-Thalassemia Major; Fetal hemoglobin; Hydroxyurea; Metformin
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Group A) Tablet Metformin (Active Comparator): Tablet Metformin 500 mg/dose orally twice a day with meal for 1 year
  Interventions: Drug: Tablet Metformin (Group A)
- (Group B) Tablet Hydroxyurea (Active Comparator): Tablet Hydroxyurea 10-20mg/kg once daily orally with breakfast for 1 year
  Interventions: Drug: Tablet Hydroxyurea (Group B)

INTERVENTIONS:
Drug: Tablet Metformin (Group A) — Tablet Metformin 500 mg/dose orally twice a day with meal for 1 year
  Other Names: Tab. Glucophage 500mg
  Arms: (Group A) Tablet Metformin
Drug: Tablet Hydroxyurea (Group B) — Tablet Hydroxyurea 10-20mg/kg once daily orally with breakfast for 1 year
  Other Names: Cap. Hydrea 500mg
  Arms: (Group B) Tablet Hydroxyurea

SUMMARY:
This clinical trial aims to evaluate and compare the effects and safety of hydroxyurea and metformin in transfusion-dependent beta-thalassemia major and correlate responders/non-responders with the single nucleotide polymorphism mutations (SNPs) by DNA analysis.

The main question to answer is:

* Is there a significant difference in the effects and safety of hydroxyurea and metformin in transfusion-dependent beta-thalassemia major?

Participants will be divided into two treatment groups. Participants of group A will receive Tab. Metformin 500mg/dose twice daily orally for one year. Participants of group B will receive Tab. Hydroxyurea 10-20mg/kg once daily orally for one year.

At the end of the study, Investigators will compare the effects and safety of hydroxyurea and metformin in transfusion-dependent beta-thalassemia major and correlate responders/non-responders with the single nucleotide polymorphism mutations (SNPs) by DNA analysis.

DETAILED DESCRIPTION:
The study will be conducted after obtaining approval from the Institutional Review Board (IRB) at Bahria University Health Sciences Campus Karachi (BUHSCK) and the Faculty Research Committee (FRC). After obtaining written informed consent, 48 participants in each group with beta-thalassemia major will be selected from the National Institute of Blood Diseases and Bone Marrow Transplantation. Participants will be randomized into two treatment groups using computer-generated randomization.

Group A participants will receive Metformin 500 mg/dose twice daily orally for one year. Group B participants will receive Hydroxyurea 10-20 mg/kg once daily orally for one year.

Dose escalation therapy will be implemented to improve participant compliance and tolerance. The first month will not be included in the study period for each participant. A general physical examination will be conducted monthly. Blood pressure (mm Hg) will be assessed using a sphygmomanometer. The pulse rate (beats per minute) will be determined by palpating the radial artery, and the Body Mass Index (kg/m^2) will be calculated for each participant.

Dietary Counseling

People with thalassemia are advised to consume vitamin C-rich foods like vegetables and fruits to prevent depletion from iron overload. They should also include dairy products in their diet to counter calcium depletion, while avoiding high-iron foods such as beef, liver, spinach, and dates.

SF (Short-form) Questionnaire

All participants will complete the SF-36, a 36-item Short-Form Health Survey, at baseline, 6 months, and 12 months. The SF-36 is a widely used tool for evaluating overall health status, consisting of 36 items across 8 domains. The scores contribute to two main components: the physical component summary (PCS) and the mental component summary (MCS). The SF-36 is employed to assess Health-Related Quality of Life (HRQoL) in both the general population and individuals with various medical conditions, including beta-thalassemia major (β-TM), allowing for comparisons of HRQoL across different illnesses and health statuses.

I) Baseline Investigations/Parameters (at day zero)

Baseline investigations will include Complete Blood Count (CBC), Random Blood Sugar (RBS), Erythrocyte Sedimentation Rate (ESR), Serum Creatinine, Serum Ferritin, Liver Function Tests (LFTs), HCV RNA test, Fetal Hemoglobin (HbF) level, Abdominal Ultrasound, Dual-Energy X-ray Absorptiometry (DEXA) Scan, and DNA mutations. Health-Related Quality of Life (HRQoL) will be assessed by the SF-36 Questionnaire at baseline, 6 months, and 12 months.

II) Monthly Follow-up for Clinical Features

Only CBC will be performed monthly, and any adverse effects related to the drugs will be inquired about.

III) At 3 Months

CBC, RBS, Serum Creatinine, and LFTs will be assessed for any adverse effects on blood, kidneys, and liver.

IV) At 6 & 12 Months

All baseline investigations, except DNA mutations, will be repeated.

V) At 9 Months

Random Blood Sugar, Serum Ferritin, and Serum Creatinine will be assessed.

Adverse Effects of Drugs

Adverse effects will be explained to each participant as follows: A) Metformin: nausea, vomiting, abdominal bloating, diarrhea, etc. B) Hydroxyurea: cytopenia, nausea, vomiting, abdominal pain, rashes, etc.

DNA mutations will be analyzed using Amplification Refractory Mutation System-Polymerase Chain Reaction (ARMS-PCR) in responders and non-responders.

Data will be collected using the Consent Form and SF-36 Questionnaire. Data analysis will be performed using IBM Statistical Package for the Social Sciences (SPSS), version 27. A p-value ≤ 0.05 will be considered statistically significant. Descriptive statistics (mean ± SD) will be used for continuous variables, while categorical variables will be presented as frequencies and percentages. To determine the mean difference, a repeated-measures two-way ANOVA within each group will be used. For correlation analysis, an independent T-test will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of beta-thalassemia major
* Transfusion dependent patients and on iron chelating agents
* Males and females 10 to 25 years of age
* Creatinine ≤1.4 mg/dL
* Written informed consent from the patients and up to 18 years consent from the Parents/Guardians.

Exclusion Criteria:

* Failure to meet inclusion criteria
* Refusal to participate
* Creatinine >1.4mg/dL
* Liver function tests (ALT and conjugated bilirubin) > 4 times upper limits of normal
* Massive splenomegaly & Liver fibrosis
* Patient on growth hormone
* Sickle beta thalassemia
* Severe osteoporosis
* Hepatitis B & C
* HIV

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-09-16 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fetal Haemoglobin (HbF) Percentage in responders and non-responders | 6 months to 1 year after the baseline
  Assessment will be done at 6 months and 1 year after the baseline
Change in frequency of blood transfusions | 6 months to 1 year after the baseline
  Assessment will be done at 6 months and 1 year after the baseline

SECONDARY OUTCOMES:
Change in quality of life assessed by the 36-Item Short Form Health Survey (SF-36) Questionnaire | 6 months to 1 year from the baseline
  Assessment will be conducted on a scoring scale of 0 to 100, with 0 being the lowest and 100 the highest possible scores, at 6 months and 1 year after the baseline.
Correlations of responders and non-responders with DNA mutations | After 1 year at the end of study
  Assessment will be done after 1 year from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Khan, MBBS MPhil, Principal Investigator — Bahria University Islamabad
Locations (1):
- Bahria University Health Sciences Campus, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD data will become accessible one year after publication and will remain available indefinitely.
Access Criteria: All the data will be accessible to everyone.

REFERENCES:
- [Background] ElTagui M, El-Ghamrawy M, AlDeeb SK, Nassim MS. Metformin as a Fetal Hemoglobin Inducer in Non-transfusion Dependent Thalassemia Patients. Indian J Hematol Blood Transfus. 2024 Jan;40(1):68-73. doi: 10.1007/s12288-023-01662-1. Epub 2023 May 5. PMID 38312174
- [Background] Yasara N, Wickramarathne N, Mettananda C, Silva I, Hameed N, Attanayaka K, Rodrigo R, Wickramasinghe N, Perera L, Manamperi A, Premawardhena A, Mettananda S. A randomised double-blind placebo-controlled clinical trial of oral hydroxyurea for transfusion-dependent beta-thalassaemia. Sci Rep. 2022 Feb 17;12(1):2752. doi: 10.1038/s41598-022-06774-8. PMID 35177777
- [Background] Arian M, Mirmohammadkhani M, Ghorbani R, Soleimani M. Health-related quality of life (HRQoL) in beta-thalassemia major (beta-TM) patients assessed by 36-item short form health survey (SF-36): a meta-analysis. Qual Life Res. 2019 Feb;28(2):321-334. doi: 10.1007/s11136-018-1986-1. Epub 2018 Sep 7. PMID 30194626
- [Background] Yasara N, Premawardhena A, Mettananda S. A comprehensive review of hydroxyurea for beta-haemoglobinopathies: the role revisited during COVID-19 pandemic. Orphanet J Rare Dis. 2021 Mar 1;16(1):114. doi: 10.1186/s13023-021-01757-w. PMID 33648529
- [Background] Mu W, Liang G, Feng Y, Jiang Y, Qu F. The Potential Therapeutic Role of Metformin in Diabetic and Non-Diabetic Bone Impairment. Pharmaceuticals (Basel). 2022 Oct 17;15(10):1274. doi: 10.3390/ph15101274. PMID 36297386
- [Background] Zhang Y, Wang H, Xiao H. Metformin Actions on the Liver: Protection Mechanisms Emerging in Hepatocytes and Immune Cells against NASH-Related HCC. Int J Mol Sci. 2021 May 9;22(9):5016. doi: 10.3390/ijms22095016. PMID 34065108
- [Background] Gluba-Brzozka A, Franczyk B, Rysz-Gorzynska M, Rokicki R, Koziarska-Rosciszewska M, Rysz J. Pathomechanisms of Immunological Disturbances in beta-Thalassemia. Int J Mol Sci. 2021 Sep 7;22(18):9677. doi: 10.3390/ijms22189677. PMID 34575839
- See also: PubMed ID: 38312174 — https://link.springer.com/article/10.1007/s12288-023-01662-1
- See also: PubMed ID: 35177777 — https://www.nature.com/articles/s41598-022-06774-8
- See also: PubMed ID: 30194626 — https://link.springer.com/article/10.1007/s11136-018-1986-1
- See also: PubMed ID: 33648529 — https://link.springer.com/article/10.1186/s13023-021-01757-w